CLINICAL TRIAL: NCT07172165
Title: A Multicenter Study to Optimize Microembolic Signal Classification Based on Double--Blind Multiparametric Assessment by Human Experts Using an Universal Graphical Interface [MESOMEGA]
Acronym: MESOMEGA
Status: Enrolling by invitation | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Sound Vascular Neurology (Unknown); RISE-Heatlh (Unknown); CRU-RISE (Unknown); University of Ostrava (Other); Maastricht University Medical Center (Other); Justus-Liebig University Gießen Medical Center (Unknown); University of Bern (Other); Centro Hospitalar De São João, E.P.E. (Other); Houston Methodist DeBakey Heart & Vascular Center (Other)
Responsible Party: Sponsor
Other Study IDs: MESOMEGA
Record Dates: First submitted 2025-06-27; First posted 2025-09-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-05

CONDITIONS: Microemboli; Stroke; Transcranial Doppler Ultrasound
Keywords: microembolic signals (MES); decision tree; stroke; microemboli; transcranial Doppler; diagnostic standard; prediction model
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transcranial Doppler clips database: Clips of MES and non-MES events. Each clip will be 20 seconds (-10 and +10 seconds in reference to the marked event). The data presented will not be modified from its original form. The final database that will be used for expert evaluation will include the necessary clips and proportions to ensure maximum reproducibility and generalization of the data. Clips will be obtained from at least 3 different types or brands of TCD machines. A single machine cannot be the source of more than 50% of the final data set. MES will be from a variety of sources including patients with atherosclerotic disease, cardioembolic stroke, or embolic stroke of unknown source.
  Interventions: Diagnostic Test: Expert double-blind evaluation

INTERVENTIONS:
Diagnostic Test: Expert double-blind evaluation — Expert reading will be using TCDPlayer and will be blinded to clinical data, source information, and other assessments. They will manually annotate six predefined signal features: characteristic audible signal increase, characteristic wave-like of raw Doppler signals, Emboli-to-Background Ratio, Emboli-to-Mirror Ratio, signal duration, and average velocity of maximum intensity. Analysis will be completed within 90 days.

SUMMARY:
Microembolic signals (MES) is a powerful predictor of future embolic events. This study aims to develop and validate a accurate model of classification of MES obtained by transcranial Doppler. monitoring of However, MES detection is technically demanding and requires expert interpretation. By providing a reproducible framework for MES interpretation, this work aims to facilitate MES integration into future clinical trials and decision-making.

DETAILED DESCRIPTION:
Rationale

The presence of microembolic signals (MES) is a powerful predictor of future embolic events. However, MES detection is technically demanding and requires expert interpretation.

Aim We aim to develop and validate a supervised prediction model for MES classification using features extracted from transcranial Doppler (TCD) signals. The model is intended to support expert consensus and enhance classification concordance by utilizing standardized, pre-specified signal features.

Sample size estimates Sample size was estimated using the pmsampsize R package. Based on five predictors, a 1:1 proportion of MES in final dataset, a maximum Nagelkerke R² of 0.75, a shrinkage factor of 90% (to minimize overfitting), and a mean absolute error in predicted probabilities ≤ 0.05, the required sample size is 850 clips. The calculations included an 80:20 training/testing split and a 10% dropout rate.

Methods and Design The "Multicenter Study to Optimize Microembolic Signal Classification Based on Double-blind Multiparametric Assessment by Human Experts Using a Universal Graphical Interface" (MESOMEGA trial) is a prospective, randomized, double-blind, diagnostic validation study. All members of World Organization of Neurosonology, their national affiliated societies, and worldwide TCD users in the medical community will be invited to submit TCD monitoring 20-second clips of presumed solid MES or non-MES high-intensity transient signals recorded using a 2 MHz transducer from the proximal middle cerebral artery. Exclusion criteria include inseparable multiple MES (e.g., curtain) or any gaseous embolic form. Each clip will be independently assessed by two randomly allocated experts. Expert reading will be using TCDPlayer and will be blinded to clinical data, source information, and other assessments. They will manually annotate six predefined signal features: characteristic audible signal increase, characteristic wave-like of raw Doppler signals, Emboli-to-Background Ratio, Emboli-to-Mirror Ratio, signal duration, and average velocity of maximum intensity. Analysis will be completed within 90 days. A supervised decision tree model will be developed on the training dataset and validation set. Performance will be assessed using stratified k-fold cross-validation, reporting accuracy, sensitivity, specificity, and area under the receiver operating characteristic curve (AUC). Following model development, a Delphi consensus process will be used to evaluate and validate model outputs, aiming for expert agreement on model acceptability and readiness for clinical application. The study will be conducted under appropriate ethical approval and in accordance with international report standards. The study will be conducted under ethical guidelines and approval.

Study Outcomes The primary outcome is the classification of clips as MES or non-MES, using expert consensus as ground truth. The model will aim for ≥ 90% classification accuracy. Secondary outcomes include model performance without auditory parameter, interrater concordance and variability, and Delphi consensus strength.

Discussion This study will assess the performance of a supervised decision tree model for MES classification and benchmark it against prior MES detection approaches. By providing a reproducible framework for MES interpretation, this work aims to facilitate MES integration into future clinical trials and decision-making.

ELIGIBILITY:
Inclusion Criteria:

MES of presumed solid form or non-MES high intensity transient signals

Obtained from on a human subject with age equal to or more than 18years old

Obtained from proximal middle cerebral artery (M1 segment)

Clip with 20 seconds duration with clearly event of interest marked using TCDPlayer

With an overall background spectrum of reasonable quality to be analyzed

Exclusion Criteria:

MES in gaseous form

Use of ultrasound contrast agent or agitated saline in the previous 24 hours

Obtained from patients with mechanical valve

Obtained from patient during any cardiac surgery or endovascular procedure1

Obtained from patient with recent severe trauma

Clips with multiples inseparable MES (e.g. curtain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clips of Transcranial Doppler monitoring either MES or non-MES high intensity transient signals (e.g. artifacts, speckle).
Sampling Method: Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Classification of each signal as MES or Non-MES | From enrollment until December of 2026
  A MES or non-MES will be considered as such the two experts agree. If the two experts do not agree, a special board (RA, WM) will decide on classification. "Recordings that remain undetermined, or those classified as undetermined by both experts, will be excluded from the primary analysis of this study. All experts will be blinded to each other, any identification tag or clinical information. We will include five predictors in the primary analysis which are: the presence of characteristic audible signal increase, characteristic wave-like raw Doppler signals, the Emboli-to-Background Ratio (EBR), Emboli-to-mirror-ratio (EMR), time length and average velocity of maximum intensity. The calculation and definition of each predictor is detailed in table 3 and in supplemental information (Proposal for a systematic analysis and reporting of microembolic signal detection of the Microembolic Signal Detection Working Groups of the World Organization of Neurosonology).

SECONDARY OUTCOMES:
Trimmed version of the model | From enrollment until December of 2026
  To compare the model performance with and without auditory parameter To compare the subgroups of exclude MES vs non-MES how model performance
Model with extra-features | From enrollment until December of 2026
  To compare the model performance with and without a derived Embolus Distance parameter as calculated by the formula: Embolus Distance (mm) = Time length x average velocity of maximum intensity
Inter-expert variability in feature extraction. | From enrollment until December of 2026
Delphi process | From enrollment until December of 2026
  Strength of the Delphi process

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine University Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Publication of protocol and associate report sheets
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Collins GS, Moons KGM, Dhiman P, Riley RD, Beam AL, Van Calster B, Ghassemi M, Liu X, Reitsma JB, van Smeden M, Boulesteix AL, Camaradou JC, Celi LA, Denaxas S, Denniston AK, Glocker B, Golub RM, Harvey H, Heinze G, Hoffman MM, Kengne AP, Lam E, Lee N, Loder EW, Maier-Hein L, Mateen BA, McCradden MD, Oakden-Rayner L, Ordish J, Parnell R, Rose S, Singh K, Wynants L, Logullo P. TRIPOD+AI statement: updated guidance for reporting clinical prediction models that use regression or machine learning methods. BMJ. 2024 Apr 16;385:e078378. doi: 10.1136/bmj-2023-078378. PMID 38626948
- [Result] Riley RD, Ensor J, Snell KIE, Harrell FE Jr, Martin GP, Reitsma JB, Moons KGM, Collins G, van Smeden M. Calculating the sample size required for developing a clinical prediction model. BMJ. 2020 Mar 18;368:m441. doi: 10.1136/bmj.m441. No abstract available. PMID 32188600
- [Result] Wong KS, Chen C, Fu J, Chang HM, Suwanwela NC, Huang YN, Han Z, Tan KS, Ratanakorn D, Chollate P, Zhao Y, Koh A, Hao Q, Markus HS; CLAIR study investigators. Clopidogrel plus aspirin versus aspirin alone for reducing embolisation in patients with acute symptomatic cerebral or carotid artery stenosis (CLAIR study): a randomised, open-label, blinded-endpoint trial. Lancet Neurol. 2010 May;9(5):489-97. doi: 10.1016/S1474-4422(10)70060-0. Epub 2010 Mar 22. PMID 20335070
- [Result] Markus HS, Droste DW, Kaps M, Larrue V, Lees KR, Siebler M, Ringelstein EB. Dual antiplatelet therapy with clopidogrel and aspirin in symptomatic carotid stenosis evaluated using doppler embolic signal detection: the Clopidogrel and Aspirin for Reduction of Emboli in Symptomatic Carotid Stenosis (CARESS) trial. Circulation. 2005 May 3;111(17):2233-40. doi: 10.1161/01.CIR.0000163561.90680.1C. Epub 2005 Apr 25. PMID 15851601
- [Result] Castro P, Ferreira J, Malojcic B, Bazadona D, Baracchini C, Pieroni A, Skoloudik D, Azevedo E, Kaps M. Detection of microemboli in patients with acute ischaemic stroke and atrial fibrillation suggests poor functional outcome. Eur Stroke J. 2024 Jun;9(2):409-417. doi: 10.1177/23969873231220508. Epub 2023 Dec 27. PMID 38149620
- [Result] Das AS, Regenhardt RW, LaRose S, Monk AD, Castro PM, Sheriff FG, Sorond FA, Vaitkevicius H. Microembolic Signals Detected by Transcranial Doppler Predict Future Stroke and Poor Outcomes. J Neuroimaging. 2020 Nov;30(6):882-889. doi: 10.1111/jon.12749. Epub 2020 Jul 10. PMID 32648610
- [Result] Sheriff F, Diz-Lopes M, Khawaja A, Sorond F, Tan CO, Azevedo E, Franceschini MA, Vaitkevicius H, Li K, Monk AD, Michaud SL, Feske SK, Castro P. Microemboli After Successful Thrombectomy Do Not Affect Outcome but Predict New Embolic Events. Stroke. 2020 Jan;51(1):154-161. doi: 10.1161/STROKEAHA.119.025856. Epub 2019 Dec 4. PMID 31795906
- [Result] Padayachee TS, Parsons S, Theobold R, Linley J, Gosling RG, Deverall PB. The detection of microemboli in the middle cerebral artery during cardiopulmonary bypass: a transcranial Doppler ultrasound investigation using membrane and bubble oxygenators. Ann Thorac Surg. 1987 Sep;44(3):298-302. doi: 10.1016/s0003-4975(10)62077-2. PMID 2957966
- [Result] Farina F, Palmieri A, Favaretto S, Viaro F, Cester G, Causin F, Baracchini C. Prognostic Role of Microembolic Signals After Endovascular Treatment in Anterior Circulation Ischemic Stroke Patients. World Neurosurg. 2018 Feb;110:e882-e889. doi: 10.1016/j.wneu.2017.11.120. Epub 2017 Nov 28. PMID 29191539
- [Result] Spencer MP, Thomas GI, Nicholls SC, Sauvage LR. Detection of middle cerebral artery emboli during carotid endarterectomy using transcranial Doppler ultrasonography. Stroke. 1990 Mar;21(3):415-23. doi: 10.1161/01.str.21.3.415. PMID 2408197